CLINICAL TRIAL: NCT04247802
Title: A Backwards Walking Programme Following Hip and Knee Arthroplasty: A Feasibility Pilot Study
Brief Title: Backwards Walking Programme Following Hip and Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PID14748; 272567 (Other: IRAS)
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Results first posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-01

CONDITIONS: Hip Osteoarthritis; Knee Osteoarthritis; Hip Arthroplasty; Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Backwards Walking (BW) programme (Experimental): This group will undertake a routine course of one to one out-patient physiotherapy which will include a BW programme. The BW programme will be prescribed by a physiotherapist and the participant will carry it out, along with other prescribed exercises, in their own home. Each participant will initially be prescribed a 5 minute BW programme to be completed once a day. The length of the BW programme and intensity will be progressed or regressed as deemed appropriate by the treating clinician with the aim for patients to achieve at least 10 minutes of BW every day of the week.
  Interventions: Other: Backwards Walking (BW) programme
- Usual Care (Active Comparator): This group will undertake a routine course of one to one out-patient physiotherapy over 12 weeks. To allow comparison between the two groups the control group will also have up to four review appointments where their home exercise programme can be progressed or regressed. The physiotherapy treatments will be not be restricted (apart from no BW programme) to allow for a pragmatic approach based on the treating clinician's clinical judgement, however their content will be recorded on treatment logs.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Backwards Walking (BW) programme — A 12 week Backwards walking programme prescribed by a registered physiotherapist and completed as part of a home exercise programme.
  Arms: Backwards Walking (BW) programme
Other: Usual Care — A 12 week physiotherapy exercise programme EXCLUDING backwards walking
  Arms: Usual Care

SUMMARY:
Backwards walking has been shown to improve balance and walking in patients who have knee Osteoarthritis. It is not known if these benefits may also be seen after surgery in patients who have had a hip or knee replacement because of Osteoarthritis. This study will look to see if it is possible to conduct a bigger study into how effective backwards walking may be after joint replacement. Patients who come to the Nuffield Orthopaedic Centre in Oxford for a hip or knee replacement will be invited. They will be placed into one of two groups at random: a group where they have a course of physiotherapy plus a backwards walking programme or a group where they have a course of physiotherapy. The physiotherapy will last for 12 weeks and those who take part will have two study assessments. The first will be before any treatment and patients will complete five measures and also be issued with a simple tick box diary to complete over the 12 weeks. The second assessment will be after the treatment and will involve the same five measures and the diaries will be collected in. Participants at this assessment will also be asked if they would like to take part in an interview for the study. This is to see what the patients thought of the study. During the study the researcher will record things such as how many patients say 'yes' to the study and how many participants drop out of the treatment, to understand if a bigger study could take place.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 65 or older.
* Participant is willing and able to give informed consent for participation in the study.
* Participants who have received a primary unilateral hip or knee arthroplasty due to osteoarthritis.

Exclusion Criteria:

* Post-operative weight bearing restrictions.
* Post-operative complications such as infection, a deep vein thrombosis or pulmonary embolism, or failure of the wound to heal.
* Inability to undertake a backwards walking programme due to conditions such as severe cardiovascular or pulmonary disease (New York Heart Association III-IV).
* Severe dementia or communication difficulties that would prevent completion of study assessments.
* Any neurological condition.
* Further planned treatment on the same or contralateral hip or knee within the next 6 months.
* Registered as visually impaired.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Batting, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (2):
- United Kingdom (2):
  - Horton General Hospital, Banbury, Oxfordshire
  - Nuffield Orthopaedic Centre, Oxford, Oxfordshire

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Backwards Walking (BW) Programme | Usual Care
Started | 33 | 30
Completed | 22 | 20
Not Completed | 11 | 10
Not completed — Withdrawal by Subject | 1 | 3
Not completed — LTFU COVID lockdown restrictions | 10 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Backwards Walking (BW) Programme | Usual Care | Total
Number analyzed (Participants) | 33 | 30 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (5.2) | 73.4 (5) | 73.0 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 22 | 47
  Male | 8 | 8 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Berg Balance Scale
Description: The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function. All the item scores are combined to make a total from a minimum of 0 to a maximum of 56. Scores between 41-56 indicate a low risk of falls, 21-40 a medium risk and, below 20 a high risk of falls.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Backwards Walking (BW) Programme | Usual Care
Number analyzed (Participants) | 22 | 20
Score on a scale | 53 (3.5) | 52.4 (4.7)

2. Secondary Outcome: Four Square Step Test
Description: The Four Square Step Test (FSST) is used to assess dynamic stability and co-ordination. It looks at the ability of the subject to step over low objects (walking sticks placed in 'plus' sign position) forward, sideways, and backward in a square pattern clockwise and anticockwise. The subject is timed completing the stepping task as fast as possible without touching the walking sticks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: second (s)
Arm/Group | Backwards Walking (BW) Programme | Usual Care
Number analyzed (Participants) | 22 | 20
second (s) | 12.8 (6.4) | 12.3 (4.9)

3. Secondary Outcome: The Two Minute Walk Test (2MWT)
Description: The Two Minute Walk Test (2MWT) is a measure of self-paced walking ability and functional capacity, particularly for those who cannot manage the longer Six Minute Walk Test (6MWT) or 12 Minute Walk Test. The participant is encouraged to walk as fast as they can, safely, without assistance for two minutes and the distance is measured in metres (m)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: metres (m)
Arm/Group | Backwards Walking (BW) Programme | Usual Care
Number analyzed (Participants) | 22 | 20
metres (m) | 123.2 (24) | 130.8 (39.3)

4. Secondary Outcome: 30 Second Sit to Stand Test
Description: The 30 Second Sit to Stand Test is a validated clinical measure of lower body strength and dynamic balance. Also known as 30 Second Chair Stand Test (30CST), the 30 Second Sit to Stand Test is designed for testing leg strength and endurance in older adults. The test measures the number of stands a person can complete in 30 seconds. The range of number of stands are from 0 to over 20.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Backwards Walking (BW) Programme | Usual Care
Number analyzed (Participants) | 22 | 20
score on a scale | 11.9 (3.4) | 11.3 (4.6)

5. Secondary Outcome: Activities-Specific Balance Confidence Scale
Description: Activities-specific balance confidence (ABC) scale is a structured questionnaire that measures an individual's confidence during ambulatory activities without falling or experiencing a sense of unsteadiness. It consists of 16 questions gauging the individual's confidence while doing specific activities. Scores range for each item from 0 (no confidence) to 100 (completely confident). For the total score all items were added together and divided by 16 to give the average. The following cut-off scores to define level of functioning among active older adults; lower than 50 %: low level of physical functioning; 50-80 %: moderate level of physical functioning; above 80 %: high level of physical functioning.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Backwards Walking (BW) Programme | Usual Care
Number analyzed (Participants) | 22 | 20
units on a scale | 88.7 (13.5) | 87.2 (15.6)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Backwards Walking (BW) Programme | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 1/22 | 0/20
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Backwards Walking (BW) Programme (N=22) | Usual Care (N=20)
Joint dislocation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Joint dislocation post operative

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/02/NCT04247802/Prot_SAP_000.pdf